CLINICAL TRIAL: NCT00079755
Title: A Phase II Multi-Dose Study of SGN-30 (Anti-CD30 mAb) in Patients With Refractory or Recurrent Hodgkin's Disease or Anaplastic Large Cell Lymphoma
Brief Title: Study of SGN-30 (Antibody) in Patients With Refractory or Recurrent Anaplastic Large Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG030-0003; NCT00107133 (obsolete NCT alias)
Record Dates: First submitted 2004-03-12; First posted 2004-03-16 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Anaplastic Large-Cell Lymphoma
Keywords: Anaplastic Large-Cell Lymphoma; Lymphoma; antigens, CD30; Monoclonal Antibody
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Lymphoma | interventions — Brentuximab Vedotin

INTERVENTIONS:
Drug: SGN-30 (anti-CD30 mAb)

SUMMARY:
To investigate safety and antitumor activity of SGN-30 in patients with Hodgkin's Disease and anaplastic large cell lymphoma (ALCL).

As of March 22, 2005, interim analysis of the Hodgkin's Disease (HD) arm has been completed per the statistical plan in the protocol. SG030-0003 is now closed to further recruitment of HD patients.

DETAILED DESCRIPTION:
SGN-30 is the chimeric form of a novel murine monoclonal antibody (mAb), AC-10, that has specificity for CD30. The CD30 antigen has a very low expression on normal cells, but is expressed on malignant cells in Hodgkins disease and anaplastic large cell lymphoma.

This study is designed to define the toxicity profile and antitumor activity of SGN-30 in patients with refractory or recurrent Hodgkin's disease and with refractory or recurrent anaplastic large cell lymphoma. Patients will receive 6 weekly intravenous (IV) infusions of SGN-30 followed by a 4 week observation period.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have refractory or recurrent HD or refractory or recurrent ALCL.
* Patients must have histologically confirmed CD30+ HD or ALCL.
* Patients must have bidimensional measurable disease on physical examination or radiologic evaluation.
* Patients must have failed systemic chemotherapy either as initial therapy for advanced disease or as salvage therapy after initial radiotherapy for early stage disease.
* Patients may have received no more than four treatments (radiation, chemotherapy, and/or biologics) prior to enrollment.
* Patients may have received no more than one stem cell transplantation.
* Patients who have undergone stem cell transplantation must have received at least one therapy post-transplantation. Patients who have not had stem cell transplantation must be considered ineligible or refuse treatment by stem cell transplantation.
* Patients must have completed radiotherapy and/or chemotherapy at least four weeks prior to enrollment. Any prior treatment with nitrogen mustard agents, melphalan, or BCNU must have been completed at least six weeks prior to enrollment.
* Patients must have an ECOG performance status of ≤ 2 and a life expectancy > three months.
* Patients must be at least 18 years of age.
* Patients must be available for periodic blood sampling, study-related assessments, and management of toxicity at the treating institution.
* Females of childbearing potential must have a negative β-HCG pregnancy test result within three days of enrollment. All patients must agree to use an effective contraceptive method during the course of the study.
* Patients must give written informed consent. A copy of the signed informed consent form will be retained in the patient's chart.
* Patients must meet baseline lab data requirements.

Exclusion Criteria:

* Patients with primary cutaneous ALCL
* Patients who have been treated previously with any anti-CD30 antibody
* Patients who have received any mAb unless a recent serum testing reveals no antibody titer and no evidence of human anti-murine antibodies (HAMA) or human anti-chimeric antibodies (HACA) in the peripheral circulation
* Patients receiving any investigational biological agent within eight weeks of enrollment or any other investigational agent within four weeks of enrollment
* Patients with a known hypersensitivity to recombinant proteins or any excipient contained in the drug formulation
* Patients with a history of other malignancies during the past five years with the exception of adequately treated basal or squamous cell skin cancer or cervical carcinoma in situ
* Patients with known active viral, bacterial, or systemic fungal infection; patients who are known to be HIV, Hepatitis B, or Hepatitis C positive.
* Patients with symptomatic cardiac disease including ventricular dysfunction, coronary artery disease, or arrhythmias
* Patients with symptomatic brain metastases requiring treatment
* Patients who are pregnant or breastfeeding
* Patients with any serious underlying medical condition that would impair their ability to receive or tolerate the planned treatment
* Patients with dementia or altered mental status that would preclude understanding and rendering of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of Califorinia at Los Angeles, Los Angeles, California
  - Georgetown University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Kaiser Permanente, Portland, Oregon
  - Oregon Health Science University, Portland, Oregon
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Result] Wahl AF, Klussman K, Thompson JD, Chen JH, Francisco LV, Risdon G, Chace DF, Siegall CB, Francisco JA. The anti-CD30 monoclonal antibody SGN-30 promotes growth arrest and DNA fragmentation in vitro and affects antitumor activity in models of Hodgkin's disease. Cancer Res. 2002 Jul 1;62(13):3736-42. PMID 12097283
- [Result] Forero-Torres A, Leonard JP, Younes A, Rosenblatt JD, Brice P, Bartlett NL, Bosly A, Pinter-Brown L, Kennedy D, Sievers EL, Gopal AK. A Phase II study of SGN-30 (anti-CD30 mAb) in Hodgkin lymphoma or systemic anaplastic large cell lymphoma. Br J Haematol. 2009 Jul;146(2):171-9. doi: 10.1111/j.1365-2141.2009.07740.x. Epub 2009 May 19. PMID 19466965
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19466965